CLINICAL TRIAL: NCT00720525
Title: Diagnostic Value of Measures of Pulsatile Versus Steady State Hemodynamics in Diastolic Heart Failure
Brief Title: Pulsatile and Steady State Hemodynamics in Diastolic Heart Failure
Status: Completed | Type: Observational
Sponsor: Klinikum Wels-Grieskirchen (Other)
Responsible Party: Dr Thomas Weber, Cardiology Department, Klinikum Wels-Grieskirchen, Austria
Other Study IDs: EK 248
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Diastolic Heart Failure
Keywords: arterial stiffness; arterial wave reflections; diastolic heart failure
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with diastolic heart failure
- 2: Patients without diastolic heart failure

SUMMARY:
Over the past few years, there has been a growing appreciation that a large number of patients with heart failure have a relatively normal (or preserved) ejection fraction (NFNEF). Epidemiologically, HFNEF is most prevalent among elderly women, most of whom have hypertension, diabetes, or both and often coronary artery disease (CAD). Increased arterial stiffness and/or wave reflections have been described in the same patient groups. Therefore, the investigators speculate that pulsatile hemodynamics, representing arterial stiffness and/or arterial wave reflections, 1) may be altered in HFNEF patients, 2) this may contribute to pathophysiology of HFNEF, and 3) this may be used for the diagnosis of the syndrome.

ELIGIBILITY:
Inclusion Criteria:

* exertional dyspnea
* undergoing heart catheterization for diagnosis or exclusion of coronary artery disease
* normal EF (> 50%)

Exclusion Criteria:

* atrial fibrillation
* more than mild valvular heart disease
* pericardial disease
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing invasive assessment for exertional dyspnea
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2008-04; Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Weber, MD, Principal Investigator — Cardiology Department, Klinikum Wels-Grieskirchen, Austria
Locations (1):
- Cardiology Department, Klinikum Wels-Grieskirchen, Wels, Austria

REFERENCES:
- [Derived] Weber T, Wassertheurer S, O'Rourke MF, Haiden A, Zweiker R, Rammer M, Hametner B, Eber B. Pulsatile hemodynamics in patients with exertional dyspnea: potentially of value in the diagnostic evaluation of suspected heart failure with preserved ejection fraction. J Am Coll Cardiol. 2013 May 7;61(18):1874-83. doi: 10.1016/j.jacc.2013.02.013. Epub 2013 Mar 6. PMID 23500307